CLINICAL TRIAL: NCT00632658
Title: Development and Validation of a Symptoms Scale for Children With Chronic Graft-versus-Host Disease
Brief Title: Development and Validation of a Symptom Scale for Children With Chronic Graft-versus-Host Disease
Acronym: cGVHD
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: University of Minnesota (Other); Dana-Farber Cancer Institute (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: SCT 0208B
Record Dates: First submitted 2008-03-04; First posted 2008-03-11 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Graft vs Host Disease
Keywords: cGVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cGVHD: Pediatric Patients with cGVHD will be asked to participate in an interview with their Physician. The interview will ask the pediatric patients questions about their cGVHD. The interview will be audio-recorded.

SUMMARY:
Chronic Graft-versus-Host Disease (cGVHD) is an important cause of morbidity and mortality in patients undergoing allogeneic bone marrow transplantation. cGVHD usually occurs after 100 days following transplantation and develops in 20-60% of transplant recipients. The incidence of cGVHD varies depending on the age of the marrow recipient, the use of sibling or unrelated donor bone marrow, the use of unmanipulated T cell-depleted bone marrow, and perhaps other factors. Clinically, cGVHD is characterized by multi-system disease, which frequently mimics the clinical features of autoimmune diseases. The manifestations include skin changes (lichenoid and sclerodermatous changes, changes in pigmentation, loss of accessory structures such as hair, dystrophic nails, and rash), joint contractures, severe cramping, hepatic dysfunctions, sicca syndrome, obstructive lung disease, esophageal dysmotility, weight loss, polyserositis, immunodeficiency, and autoantibodies including anti-nuclear antibody, anti-erythrocyte antibodies, and anti-platelet antibodies.

DETAILED DESCRIPTION:
A large number of children with cGVHD have to deal with many years of a disfiguring and painful chronic illness with the side effects of long term steroid use. The number of stem cell transplants done in children is only growing given that we are now transplanting patients with a variety of nonmalignant disorders and given the use of alternative donor sources. The broad categories of limited and extensive cGVHD are recognized by clinicians, but are not particularly useful in clinical practice. Since cGVHD may involve almost every organ system adn since cGVHD constitutes a waxing and waning nature, cGVHD makes clinical management very difficult and complicated. Currently, there is a symptoms scale used in the adult population for measuring symptom burden for adults with cGVHD. This scale is called the "Lee Symptoms Scale". The purpose of this project is to develop a scale that is similar in design to the Lee Scale, but it is specifically designed to measure the burden of cGVHD in the pediatric population

ELIGIBILITY:
Inclusion Criteria:

* 5-18 years of age
* Prior allogeneic Stem Cell Transplant, with any graft source, donor type, and GVHD prophylaxis allowed
* Clinical diagnosis of cGVHD
* Need for systemic treatment, defined as any medication or intervention delivered
* No evidence of primary disease relapse
* Signed, informed consent, and if applicable, adolescent assent

Exclusion Criteria:

* Inability to give signed informed consent

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with cGVHD will be identified by their local physican and asked to participate in this research study. A total of 24 children will be asked to participate in this study. The parents of all of the 24 children will also be asked to participate and give us their feed-back on what it is like to cope with a child with cGVHD.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To develop a Pediatric Chronic GVHD Symptoms Scale (PCSS) that reliably measures the disease specific burden of chronic GVHD in children | One Day Interview will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Reggie E Duerst, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States